CLINICAL TRIAL: NCT03384706
Title: A Comparison of Cognitive Processing Therapy (CPT) Versus Accelerated Resolution Therapy (ART) Versus Wait List (WL)
Brief Title: A Comparison of CPT Versus ART Versus WL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Cincinnati VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Chard, Director, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1590
Record Dates: First submitted 2017-07-20; First posted 2017-12-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder (PTSD); Clinical Trial; Psychotherapy; Assessment; Effectiveness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study will examine the effectiveness of Cognitive Processing Therapy (CPT) as compared to Accelerated Resolution Therapy (ART) and a Waitlist (WL) control using a Randomized, Cross-Over Design. 280 participants will be randomly assigned to ART, CPT or WL. Upon completion of the WL condition, participants will be re-randomized to ART or CPT.
Who Masked: Outcomes Assessor
Masking Description: The assessors will remain blind to treatment condition throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Processing Therapy (CPT) (Active Comparator): PTSD Psychotherapy CPT will be implemented using the Cognitive-Only version, excluding the trauma account.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)
- Accelerated Resolution Therapy (ART) (Experimental): PTSD Psychotherapy
  Interventions: Behavioral: Accelerated Resolution Therapy (ART)
- Wait List Control (No Intervention): Wait List control will include a 7 week minimal attention control period with weekly check-in calls to ensure that the participant has not experienced any significant worsening in their symptoms that might require interventions, (e.g. suicidal intent).

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — CPT looks at the impact the traumatic event has had on your life and helps you to examine and change unhelpful thoughts and feelings related to the event, yourself, others and the world.
  CPT will be conducted in 5-15, 60 minute sessions held once or twice a week.
  Arms: Cognitive Processing Therapy (CPT)
Behavioral: Accelerated Resolution Therapy (ART) — ART, like CPT also involves processing thoughts and feelings related to the event, but does this in a different way relying more on visualization or imagination rather than talking.
  ART will be conducted in 5-15, 60 minute sessions held once or twice a week.
  Arms: Accelerated Resolution Therapy (ART)

SUMMARY:
The purpose of this research study is to compare the effectiveness of two treatments for the symptoms of Posttraumatic Stress Disorder (PTSD) with a no therapy, wait-list control condition. The two treatments are Cognitive Processing Therapy (CPT) as compared to Accelerated Resolution Therapy (ART). Both have been found to be effective with veterans and civilians in prior studies but they have never been compared to one another. Participants will be 280 males and females ages 18 and older who meet criteria for PTSD (or subthreshold PTSD). PTSD is a condition that can occur after a trauma experience such as combat, sexual abuse, physical abuse, or natural disasters.

DETAILED DESCRIPTION:
Objective(s): The primary aim of this study is to examine the effectiveness of two treatments for the symptoms of Posttraumatic Stress Disorder (PTSD) with a no therapy, wait list control condition. The two treatments are Cognitive Processing Therapy (CPT) as compared to Accelerated Resolution Therapy (ART). Additional related symptoms of depression, anger, sleep, and physical health will also be assessed. The study will involve both civilians and veterans seeking outpatient therapy for PTSD. Data will be obtained via clinician structured interviews and self-report measures.

Research Design: Participants will be recruited from the Cincinnati VA Medical Center, Trauma Recovery Center (TRC), and at the University of Cincinnati (UC) Health Stress Center located in Cincinnati, Ohio. All eligible participants will be randomized to receive CPT, ART, or Wait List (WL) condition. For participants who are randomized to the WL condition, following a period of seven weeks will be randomized into one of the two active treatment conditions, CPT or ART. Participants in the two active treatment conditions will complete an assessment at pre-treatment, post-treatment, 3 month, and 1 year follow-up.

Methodology: Participants will include 280 males and females ages 18 and older who meet criteria for PTSD (or subthreshold PTSD). The investigators will contact potential participants to determine eligibility for the study assessing inclusionary and exclusionary criteria. All eligible participants will then be asked to complete a pre-treatment assessment prior to being assigned their study treatment (CPT or ART or WL). Participants will receive a full course of outpatient CPT or ART depending on their assigned study treatment. Once the participant and treating clinician determine that therapy has been fully completed, participants will complete a post-treatment assessment. Follow-up assessments will then be completed 3-months and 1-year following the completion of therapy.

At each assessment participants will be asked to complete a series of self- and clinic-reported measures that include assessments of PTSD symptoms, depression, general mental health, pain, sleep habits, and health care utilization.

Findings: Not applicable at this time.

Clinical Relationships: The investigators anticipate that understanding the comparative effectiveness between CPT and ART therapies will provide necessary information for care provided to civilians and veterans suffering from PTSD.

ELIGIBILITY:
Inclusion Criteria:

* May have posttraumatic stress disorder (PTSD)

Exclusion Criteria:

* Meet criteria for unmedicated bipolar, mania, or unmedicated psychotic disorders
* Meet criteria for a substance use disorder requiring detoxification treatment
* Have active suicidal or homicidal intent with (a) plan(s) and (a) means
* Have a medical condition that will interfere with twice weekly therapy sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity | Through study completion, an average of 15 months
  Combined Clinician-Administered PTSD Scale for DSM-IV and DSM-5 (CAPS-IV/CAPS-V)

SECONDARY OUTCOMES:
Depression symptom severity | Through study completion, an average of 15 months
  Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Chard, PhD, Principal Investigator — Cincinnati VA Medical Center; University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati VA Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03384706/Prot_SAP_000.pdf